CLINICAL TRIAL: NCT01101217
Title: Effect of Zinc Suplementation on Serum Hemosystein Level in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Office of Vice Chancellor for research in Shiraz UMS, Shiraz University of Medical Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4542
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2009-01

CONDITIONS: End Stage Renal Failure
Keywords: hemocystein zinc renal failure
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): placebo for 6 weeks
  Interventions: Drug: placebo
- zinc (Active Comparator): zinc sulfate 220 mg per day orally for 6 weeks
  Interventions: Drug: Zinc Supplement

INTERVENTIONS:
Drug: Zinc Supplement — in 50 patients zinc sulfate 220 mg per day orally for 6 weeks
  Arms: zinc
Drug: placebo — placebo daily for 6 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to study the effect of zinc supplementation in end stage renal failure on hemocystein level.

DETAILED DESCRIPTION:
hemocystein increased in end stage renal failure and zinc involved in hemocystein metabolism thus zinc supplementation may be effective on hemocystein level.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis for 3 months
* older than 18 years old
* serum level of zinc less than 72.6 microgram/ l in men and less than 70 microgram/ l in female

Exclusion Criteria:

* acute renal failre
* malabsorption
* history of steroid or cytotoxic consumption

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
decreased hemocystein level | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University Hemodialysis Center, Shiraz, Fars, Iran